CLINICAL TRIAL: NCT05005806
Title: Randomised Double-blind Placebo-controlled Clinical Trial of Fish Oil (Omega 3 ) in Sjögren's Syndrome Patients
Brief Title: Fish Oil (Omega 3 ) in Sjogren's Syndrome
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hawler Medical University (Other)
Responsible Party: Principal Investigator, Aryan Mohamadfatih Jalal, principal investigator, Hawler Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Fish oil in Sjogren Syndrome
Record Dates: First submitted 2021-08-05; First posted 2021-08-16 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2022-04

CONDITIONS: Sjogren's Syndrome
Keywords: Sjogren's syndrome; Omega 3 fatty acid; dry eye; dry mouth
MeSH Terms: conditions — Sjogren's Syndrome; Dry Eye Syndromes; Xerostomia | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Intervention Model Description: 100 participants will asses for eligibility and underwent randomized double blind placebo controlled clinical trial .in whom they meet inclusion criteria with informed consent from participants and will be held at out patient clinic of Rheumatology department at Erbil- Iraq.
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omega 3 soft gel (Active Comparator): participants in this group (1)omega 3 fatty acid soft gel 1000 mg will be given to participants twice daily for two months.
  Interventions: Drug: Omega 3 fatty acid
- placebo (Placebo Comparator): placebo group ,placebo soft gel designed same as omega 3 contain Vitamin A 1000 mg twice daily for two months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Omega 3 fatty acid — omega 3 fatty acid soft gel
  Arms: Omega 3 soft gel
Drug: Placebo — placebo soft gel
  Arms: placebo

SUMMARY:
Sjögren's syndrome (pSS) is an autoimmune disorder affecting mainly the exocrine glands.this lead to dryness of the main mucosal surface ,such as the mouth ,eye,skin nose,pharynx,larynx and vagina . The history of the disease is characterized by a slowly progression of sicca symptoms and fatigue; however, a subset of patients would experience extra glandular activity. Lipid mediators derived from polyunsaturated fatty acids, related to inflammation and immune response regulation. In this sense, the polyunsaturated fatty acids omega-3 (ω-3 FA) have been associated with several illnesses such as cancer, cardiovascular disease and autoimmune diseases and their balance at the cellular membranes can result in an anti-inflammatory .

DETAILED DESCRIPTION:
this is a randomized double -blind placebo -controlled clinical trial .the participants will be randomize into two groups .Group 1 receive dietary omega-3 supplementation (omega-3 group) whereas Group 2(placebo group) receive a placebo . The two types are similar to each other in the form of soft gel ,both are given two times daily for two months with follow-up of patients whom they full fill the inclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Age≥ 18 and ≤ 70 years old .
* Able to provide inform consent
* Patients diagnosed as syndrome according to 2016 ACR(American college of Rheumatology)/ EULAR(European league Against Rheumatism classification criteria for Sjögren's syndrome

Exclusion Criteria:

* any preexisting ocular disease or on eye drops lubricants.
* patients on (Beta blockers, Diuretics , anticholinergic, α 1antagonist and α 2 agonist ,anticoagulant, antidepressant, antihistamine ,pilocarpine, cevimeline ) .
* past history of diabetes, psychiatric disorder.
* pregnancy, lactating mother
* malignancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-09-02 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-07 (Actual)

PRIMARY OUTCOMES:
Dry eye symptoms | up to two months
  subjective symptoms of dry eye which involve 6 symptoms( burning sensation, itching, foreign body sensation , Dryness, mucous discharge, photophobia) when absent(0) , sometime present (1) , frequently present (2), always present (3) ( score 0-6 mild, 6-12 moderate, 12-18 sever by visual analogue scale
Dry mouth symptoms | up to two months
  measure dry mouth by inventory xerostomia score is included 11 questionnaire which score calculated by visual analogue scale from 1 to 5 ( never to very often ) have symptoms

SECONDARY OUTCOMES:
schirmers tear test | up to two months
  patient will sitt in examining chair ,the test strip is bend with round wick and at indentation ( approximately 90 degree ) then patient instruct to look up and draw eye gently downward ,then round bend end of sterile strip hook over eyelid border at junction of middle and outer one third of the lower eyelid margin.
sialometry test | up to two months
  measuring of salivary flow ,unstimulated whole saliva is collect when mouth rinse with distill water then the patient tow his head and try not to move during the test, a plastic disposable pipette drew the accumulated saliva in the floor of the mouth,for a period of five minute,the volume will record ,flow express as ml/min.

CONTACTS AND LOCATIONS:
Overall Officials: Ziad SH AL Rawi, F R C P London, Study Director — Professor of Rheumatolgy,Baghdad University; Aryan MF Jalal, M.B.CH.B, Principal Investigator — Rheumatology,Hawler medical uiversity,Kurdistan Board for medical specialities; Ibtihal HH Faraj, M-B.CH.B, Principal Investigator — Rheumatology,Hawler medical university
Locations (1):
- Reumatology out patient clinic,, Erbil, Iraq